CLINICAL TRIAL: NCT04819607
Title: The Evaluating Multidisciplinary Bone Marrow Failure Care in Bone Marrow Failure and Related Disorders.(The EMBRACE Study)
Brief Title: The Evaluating Multidisciplinary Bone Marrow Failure Care in Bone Marrow Failure and Related Disorders.
Acronym: EMBRACE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Other Study IDs: 21/44
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Bone Marrow Failure Syndrome; Aplastic Anemia
MeSH Terms: conditions — Bone Marrow Failure Disorders; Anemia, Aplastic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BMFS patients: Patients with BMFS attending Peter MacCallum Cancer Centre haematology clinic.
  Interventions: Other: model of care

INTERVENTIONS:
Other: model of care — Multidisciplinary model of care for BMFS patients.

SUMMARY:
This is a prospective hybrid implementation-effectiveness study of a model of care for patients with bone marrow failure syndromes and inherited predisposition to haematological malignancy that includes comprehensive diagnostic genomic evaluation, multidisciplinary case review, provision of clinical care including from clinical haematologists, medical geneticists and genetic counsellors.

DETAILED DESCRIPTION:
The inherited bone marrow disorders (IBMD) comprise both the traditional inherited bone marrow failure syndromes (BMFS) and the more recently described entity of germline predisposition to haematological malignancy. Patients with IBMD often present highly complex health issues that are unique and not commonly encountered. As a consequence, clinicians may feel less confident in managing these unique issues given their lack of frequent exposure to this patient group. Recent advances in genomics have resulted in more accurate diagnosis of IBMD and their subtyping and have resulted in a rapidly evolving field with multiple opportunities to improve patient outcomes.

Stage 1 of this study evaluated and quantified the current challenges faced by 3 stakeholder groups, patients with IBMD, patient advocates and nationally, clinicians who care for IBMD patients. The results demonstrated that the challenges described in Stage 1 may be overcome by instigating a multidisciplinary approach to care for BMF patients. Interventions designed to address the challenges identified in stage 1 form the model of multidisciplinary care to be implemented in the Peter MacCallum Cancer Centre/ Royal Melbourne Hospital clinic. The model of care involves:

1. Provide access to genetic testing with expert result interpretation
2. Presentation of clinical information and relevant investigations (including genetic) at a multidisciplinary team meeting involving haematologists, molecular haematopathologists, clinical genetics, genetic counsellors, scientists and specialised nurses.
3. Provision of a suggested care plan to clinician
4. Genetic counselling and provision of written disease specific information including details of suggested care plan to patient
5. Genetic counselling and provision of written information and access to testing for at risk family members
6. Dedicated team focused on many individually rare diseases with a demonstrated focus on provision of comprehensive care
7. Opportunity to participate in local and international research

The EMBRACE study will focus on evaluating the model of care.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following criteria for study entry:

1. Age > or = 18 years at enrolment
2. Able to give informed consent (or responsible family member able to give informed consent)
3. Patient is receiving care under the institutional guidelines/stream model of care

Exclusion Criteria:

1. Patient not eligible for management under the model of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of inherited bone marrow disorder (IBMD) including traditional inherited bone marrow failure syndromes (BMFS) and germline predisposition to haematological malignancy who meet all the inclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
to assess the effectiveness and implementation of the model of care through a mixture of objective metrics and patient /physician reported outcomes | 12 months
  Effectiveness - patient/physician reported outcomes of satisfaction with model of care as measured by questionnaire Implementation - compliance with of model as measured by audit against pre-specified key performance indicators

SECONDARY OUTCOMES:
To assess longitudinal quality of life assessment in patients being treated with the model | 12 months
  Longitudinal quality of life assessment in patients being treated with the model measured by the EORTC QLQ-C30
To quantitate healthcare usage of patients within the model | 12 months
  Quantitate healthcare usage of patients within the model measured by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Piers Blombery, MBBS(Hons), Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No